CLINICAL TRIAL: NCT02658942
Title: Flexible Ureteroscopy Versus ESWL in the Management of Lower Calyceal Stones: A Prospective Randomized Study
Brief Title: Flexible Ureteroscopy Versus ESWL in the Management of Lower Calyceal Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohammed said elsheemy, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 62120
Record Dates: First submitted 2016-01-14; First posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Renal Stones
Keywords: renal stones; lower calyx; Ureteroscopy; Shockwave lithotripsy; Holmium laser; Adult; Kidney
MeSH Terms: conditions — Nephrolithiasis | interventions — Ureteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ureteroscopy (Active Comparator): Intervention: Flexible ureteroscopy for removal of lower calyceal stones using holmium:YAG laser lithotripsy
  Interventions: Procedure: Ureteroscopy
- Shockwave lithotripsy (Active Comparator): Intervention: Shockwave lithotripsy for lithotripsy of lower calyceal stones using Siemens Lithostar Lithotriptor
  Interventions: Procedure: Shockwave lithotripsy

INTERVENTIONS:
Procedure: Ureteroscopy — In Group A patients, Karl Storz Flex-X 7.5, FURS with a 365 µm laser fiber.
  Other Names: Flexible Ureteroscopy
  Arms: Ureteroscopy
Procedure: Shockwave lithotripsy — In Group B patients, a Siemens Lithostar Lithotriptor
  Other Names: ESWL
  Arms: Shockwave lithotripsy

SUMMARY:
to assess safety, efficacy of Flexible ureteroscopy (FURS) holmium:YAG laser lithotripsy (LL) compared to extracorporeal shockwave lithotripsy (ESWL) in management of lower calyceal stones (LC) stones.

DETAILED DESCRIPTION:
to assess stone free rate, number of sessions and complications of flexible ureteroscopy holmium:YAG laser lithotripsy compared to extracorporeal shockwave lithotripsy in the management of lower calyceal stones less than 2 cm in size.

ELIGIBILITY:
Inclusion Criteria:

* unilateral
* radiopaque stone(s)
* < 2 cm
* located in the lower calyx.

Exclusion Criteria:

* Bleeding tendency
* distal obstruction
* Anomalies of the urinary tract
* Solitary kidney

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Stone free rate | 3 months
  no stone fragments or having fragments <3mm

SECONDARY OUTCOMES:
Complications | 3 years
  Bleeding Infection Pain obstruction renal or ureteric injury UTI Fever

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed S ElSheemy, M.D, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt